CLINICAL TRIAL: NCT05188079
Title: Effect of Acute Nitrate Supplementation on Vascular Function in Hispanic, Black and White Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY00001163
Record Dates: First submitted 2021-12-08; First posted 2022-01-12 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Healthy Adults

STUDY DESIGN:
Intervention Model Description: randomized, cross-over, placebo-controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: it will be double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beetroot Juice (Active Comparator): 140 ml of beetroot juice (high nitrate dietary supplement)
  Interventions: Dietary Supplement: Beetroot juice
- Placebo (Placebo Comparator): Placebo drink looks and tastes like the beetroot juice but has the nitrate removed from the juice.
  Interventions: Dietary Supplement: Placebo drink

INTERVENTIONS:
Dietary Supplement: Beetroot juice — high nitrate supplement
  Arms: Beetroot Juice
Dietary Supplement: Placebo drink — placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess vascular function in African Americans, Hispanic and Caucasian Americans to better understand racial differences in cardiovascular health. The investigators will further investigate the affect of Beetroot juice on the vascular function of all participants.

DETAILED DESCRIPTION:
African Americans and Hispanic individuals have the highest incidence of type 2 diabetes, which increases their risk of all cardiovascular diseases. One of the hallmarks of type 2 diabetes is vascular dysfunction, caused by a lack of nitric oxide bioavailability. Vascular function and blood flow responses to exercise have been shown to improve after nitrate supplementation (beetroot juice), However, whether nitrate supplementation will improve vascular function in African American and Hispanic individuals remains unknown. The investigators will perform a randomized, placebo-controlled study in healthy African American, Hispanic and Caucasian subjects. They will be studied before and 90 minutes after consuming Beetroot juice (high nitrate supplement) or Placebo, with at least 1-week washout period between the two visits (Kenjale AA et al., J Appl Physiol 2011).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women who are either Caucasian American, Hispanic, or non-Hispanic African American

Exclusion Criteria:

* Blood pressure higher than or equal to 140/90 mmHg
* BMI > 35kg/m2
* Have a history of cardiovascular, neurological or vascular diseases
* Take prescription medications
* Are smokers
* Are pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Forearm blood flow | through study completion, an average of 2 year
  Blood flow of the brachial artery will be measured continuously at rest, during 3 min of handgrip exercise and for up to 1 min after the cessation of handgrip exercise.

SECONDARY OUTCOMES:
Flow mediated vasodilation | through study completion, an average of 2 year
  The subjects will lay supine with arm extended on a side table. Resting brachial artery diameter and velocity will be measured at rest for 2 min. Following this, a pneumatic cuff will be inflated on the forearm to supersystolic pressure (220-240 Torr) for 5 min and once the cuff is released, brachial artery diameter and velocity will be measured for up to 3 minutes after cuff deflation. FMD% will be calculated as (highest diameter after cuff deflation - baseline brachial artery diameter)/ baseline diameter * 100

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin, Austin, Texas, United States